CLINICAL TRIAL: NCT05998447
Title: A Phase II Study to Evaluate the Safety and the Efficacy of GEN-001 in Combination With Pembrolizumab for Patients With Advanced Refractory Biliary Tract Cancer
Brief Title: GEN-001 Plus Pembrolizumab for Patients With Advanced Refractory Biliary Tract Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Genome & Company (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [GNC] GEN001-202; KEYNOTE-D86 (Other: Merck Sharp & Dohme LLC); MK-3475-D86 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-08-01; First posted 2023-08-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEN-001 with pembrolizumab or GEN-001 with pembrolizumab and mFOLFOX (Experimental): Drug: GEN-001
  Drug: pembrolizumab
  Drug: mFOLFOX
  Interventions: Drug: GEN-001; Drug: Pembrolizumab; Drug: mFOLFOX

INTERVENTIONS:
Drug: GEN-001 — The capsules taken by mouth. Each capsule will contain ≥ 3x10^11 colony-forming units (CFU)
Drug: Pembrolizumab — 200 mg given by intravenous (IV) infusion once every 3 weeks
  Other Names: KEYTRUDA®
Drug: mFOLFOX — mFOLFOX given by intravenous (IV) once every 2 weeks for only cohort 3

SUMMARY:
This is a phase II, multicenter, open-label study with a safety run-in to evaluate the safety and efficacy of GEN-001 in combination with pembrolizumab or in combination with pembrolizumab and mFOLFOX for patients with advanced refractory BTC who have progressed after 1 or 2 prior standard therapy and are not candidates for any other standard therapy. The safety run-in phase will be conducted before the main study phase

ELIGIBILITY:
Inclusion Criteria:

* The patient (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Be ≥19 years of age on day of signing informed consent.
* Patient with histologically or cytologically confirmed diagnosis of unresectable, recurrent, or metastatic advanced biliary tract adenocarcinoma of the gallbladder or biliary tree (either intrahepatic or extrahepatic cholangiocarcinoma)

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test (within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (Cohort 1 only), and was discontinued from the previous IO therapy due to a Grade 3 or higher immune-related AE (irAE) (Cohort 2 and Cohort 3).
* Is currently participating and receiving study treatments or has participated in a study of an investigational agent and received the study therapy or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has had an allogeneic tissue/solid organ transplan

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
The recommended Phase 2 dose (RP2D) of GEN-001 in patients with advanced refractory biliary tract cancer (BTC), when administered as combined with pembrolizumab or as combined with pembrolizumab and mFOLFOX. | 1 years
  Incidence of dose-limiting toxicity (DLT)
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by the Investigator. | 1 years
  The assessment of the anti-tumor activity per cohort

SECONDARY OUTCOMES:
Incidence of Adverse Event (AE)s and laboratory abnormalities per National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) v.5.0. cohort. | 1 years
  The assessment the overall safety and tolerability per cohort.
Duration of Response (DoR) | 1 years
  the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first
Progression-free Survival (PFS) | 1 years
  the time from the start date of treatment to the date of PD by RECIST v1.1 or death due to any cause, whichever occurs first
Overall Survival (OS) | 1 years
  the time from the start date of treatment to the date of death

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Seoul National University Hospital, Seoul, Seoul
  - Severance Hospital, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul
  - Samsung Medical Center., Seoul, Seoul
  - Korea University Guro Hospital, Seoul, Seoul
  - Ajou University Medical Center, Suwon

IPD SHARING:
Plan to Share IPD: No